CLINICAL TRIAL: NCT01452334
Title: A Phase I Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Immunoregulatory Activity, and Preliminary Antitumor Activity of Anti-Programmed-Death-Ligand 1 (PD-L1) Antibody (BMS-936559) in Subjects With Relapsed or Refractory Hematologic Malignancy
Brief Title: Safety Study of Anti-Programmed Death-Ligand 1 in Hematologic Malignancy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA210-003
Record Dates: First submitted 2011-10-04; First posted 2011-10-14 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin Lymphoma; Multiple Myeloma; Chronic Myelogenous Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — BMS-936559

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: BMS-936559 (Experimental)
  Interventions: Biological: BMS-936559 (Anti PD-L1)

INTERVENTIONS:
Biological: BMS-936559 (Anti PD-L1) — Injection for infusion, Intravenous (IV), 1, 3 or 10 mg/kg, Every 2 weeks, 48-96 weeks depending on response

SUMMARY:
The purpose of this study is to determine the side effects of treatment with the monoclonal antibody anti-PD-L1 (BMS-936559) in subjects with compromised bone marrow function and the dose that should be recommended for use in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance of 0 or 1
* Subjects must have histological confirmation of relapsed or refractory hematologic malignancy
* Subjects with non-Hodgkin's lymphoma or Hodgkin lymphoma must have at least one measureable lesion as defined by lymphoma response criteria. Tumor sites that are considered measureable must not have received prior radiation therapy
* Subjects with multiple myeloma (MM) must have detectable disease as measured by presence of monoclonal immunoglobulin protein in a serum electrophoresis: IgG, IgA, IgM, (M-protein ≥ 0.5 g/dl or serum IgD M-protein ≥ 0.05 g/dl) or serum free-light chain or 24 hour urine with free light chain. Excluded are subjects with only plasmacytomas, plasma cell leukemia, or non-secretory myeloma
* Subjects with chronic myelogenous leukemia (CML) must have evidence of the Philadelphia chromosome by polymerase chain reaction (PCR) or chromosome analysis
* Life expectancy of at least 3 months
* For subjects with lymphoma, either a formalin fixed tissue block or 7 to 15 slides of tumor sample (archival or fresh) must be available for performance of correlative studies
* Subjects must have received at least one prior chemotherapy regimen. Subjects must be off therapy for at least 4 weeks ( 2 weeks for oral agents) prior to Day 1
* Prior palliative radiation must have been completed at least 2 weeks prior to study Day 1
* Toxicities related to prior therapy must have returned to Grade 1 or less, except for alopecia. Peripheral neuropathy must be Grade 2 or less
* Adequate bone marrow function defined as:

  1. Absolute neutrophil count ≥ 1000/μl (stable off any growth factor within 1 week of study drug administration)
  2. Hemoglobin ≥ 9 g/dL (transfusion to achieve this level is permitted)
  3. Platelet count ≥ 50 X 103/ μl (transfusion to achieve this level is not permitted)
* Adequate renal parameters defined as Creatinine clearance (CrCl) > 40 ml/min (Cockcroft-Gault formula)
* Adequate hepatic parameters defined as:

  1. Aspartate aminotransferase (AST) ≤ 3 x ULN
  2. Alanine aminotransferase (ALT) ≤ 3 x ULN
  3. Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert's Syndrome, who must have total bilirubin < 3.0 mg/dL and direct bilirubin < 0.5 mg/dL)
* Women of child bearing potential (WOCBP) and for at least 70 days after the last dose of investigational product
* Men and women ≥ 18 years of age

Exclusion Criteria:

* Subjects with acute leukemias, blast phase CML, T cell lymphoblastic or Burkitt lymphoma
* Subjects with a history of central nervous system involvement by hematologic malignancy or symptoms suggestive of central nervous system involvement
* Subjects with concomitant second malignancies (except adequately treated nonmelanomatous skin cancers, ductal carcinoma in situ, treated superficial bladder cancer or prostate cancer or in situ cervical cancers) are excluded unless a complete remission was achieved at least 3 years prior to study entry and no additional therapy is required or anticipated to be required during the study period
* Subjects with any active autoimmune disease or a history of known or suspected autoimmune disease, or history of syndrome that requires systemic corticosteroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy
* A serious uncontrolled medical disorder or active infection which would impair the ability of the subject to receive protocol therapy or whose control may be jeopardized by the complications of this therapy
* Prior therapy with an anti programmed death-1 (anti-PD-1), anti Programmed death ligand 1 (anti-PD-L1), anti Programmed death ligand 2 (anti-PD-L2), anti-CD137 or anti Cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4) antibody (or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways)
* Non-oncology vaccine therapies for prevention of infectious diseases (eg seasonal flu vaccine, Human Papilloma Virus (HPV) vaccine) within 4 weeks of study drug administration Vaccination while on study is also prohibited except for administration of the inactivated influenza vaccine
* Prior organ allograft or allogeneic bone marrow transplantation
* Positive for human immunodeficiency virus (HIV 1/2) or known acquired immunodeficiency syndrome (AIDS)
* Positive tests for hepatitis B virus surface antigen (HBsAg), or antibody to hepatitis B core Ag or hepatitis C virus antibody (confirmed by Western Blot) or hepatitis C ribonucleic acid (RNA) in serum
* Ejection fraction less than 45% in subjects with prior anthracycline exposure
* History of Grade 4 anaphylactic reaction to monoclonal antibody therapy
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of BMS-936559 as measured by the incidence of adverse events (AEs), serious AEs, dose-limiting toxicities, laboratory test abnormalities, and changes in vital signs | Weeks 1
Safety and tolerability of BMS-936559 as measured by the incidence of adverse events (AEs), serious AEs, dose-limiting toxicities, laboratory test abnormalities, and changes in vital signs | Weeks 2
Safety and tolerability of BMS-936559 as measured by the incidence of adverse events (AEs), serious AEs, dose-limiting toxicities, laboratory test abnormalities, and changes in vital signs | Weeks 3
Safety and tolerability of BMS-936559 as measured by the incidence of adverse events (AEs), serious AEs, dose-limiting toxicities, laboratory test abnormalities, and changes in vital signs | Weeks 6
Safety and tolerability of BMS-936559 as measured by the incidence of adverse events (AEs), serious AEs, dose-limiting toxicities, laboratory test abnormalities, and changes in vital signs | Every 2 weeks until 70 days after last treatment

SECONDARY OUTCOMES:
Pharmacokinetics of BMS-936559 as measured by maximum observed serum concentration (Cmax) | Within the first 22 weeks, weeks 34, weeks 46, and at follow-up (35 ± 7 days after last treatment and 70-90 days since last treatment)
Pharmacokinetics of BMS-936559 as measured by time of maximum observed serum concentration (Tmax) | Within the first 22 weeks, weeks 34, weeks 46, and at follow-up (35 ± 7 days after last treatment and 70-90 days since last treatment)
Pharmacokinetics of BMS-936559 as measured by area under the serum concentration time curve in the dosing interval [AUC(TAU)] | Within the first 22 weeks, weeks 34, weeks 46, and at follow-up (35 ± 7 days after last treatment and 70-90 days since last treatment)
Pharmacokinetics of BMS-936559 as measured by accumulation index (AI) calculated ar ratio of the AUC(TAU) at steady state and first dose | Within the first 22 weeks, weeks 34, weeks 46, and at follow-up (35 ± 7 days after last treatment and 70-90 days since last treatment)
Pharmacokinetics of BMS-936559 as measured by serum concentration achieved at the end of dosing interval (trough concentration) (Cmin) | Within the first 22 weeks, weeks 34, weeks 46, and at follow-up (35 ± 7 days after last treatment and 70-90 days since last treatment)
Pharmacokinetics of BMS-936559 as measured by serum concentration achieved at the end of the infusion (Ceoinf) | Within the first 22 weeks, weeks 34, weeks 46, and at follow-up (35 ± 7 days after last treatment and 70-90 days since last treatment)
Antitumor activity of BMS-936559 as measured by the objective response rate, duration of response, and progression free survival | Week 4, week 12, week 20, and every 16 weeks until confirmed disease progression assessed up to Week 214
Immunogenicity of BMS-936559 as measured by the frequency of subjects with an increase in anti-drug antibody levels from baseline | Baseline, weeks 3, weeks 12, weeks 20, weeks 34, weeks 46, and at follow-up (35 ± 7 days after last treatment and 70-90 days since last treatment)
Programmed death ligand 1 (PD-L1) receptor occupancy levels as measured by changes from baseline | Baseline and within the first 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb